CLINICAL TRIAL: NCT02369146
Title: A Phase II, Open-label, Multiple-dose Trial to Investigate the Safety and Efficacy of UB-421 Monotherapy in Substitution for Stable Antiretroviral Therapy in HIV Infected Adults
Brief Title: To Investigate the Safety and Efficacy of UB-421 Monotherapy in HIV Infected Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: United BioPharma (Industry)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); Kaohsiung Veterans General Hospital. (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UBP-A202-HIV
Record Dates: First submitted 2015-02-05; First posted 2015-02-23 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — UB-421

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cohort 1 (Experimental): Subjects will receive 8 doses of the UB-421 by intravenous infusion at 10 mg/kg weekly
  Interventions: Drug: UB-421
- cohort 2 (Experimental): Subjects will receive 8 doses of the UB-421 by intravenous infusion at 25 mg/kg weekly
  Interventions: Drug: UB-421

INTERVENTIONS:
Drug: UB-421 — The UB-421 (dB4C7 mAb) will be supplied at a concentration of 10 mg/mL (100 mg in 10 mL vial). Subjects will receive 8 doses of the UB-421 by intravenous infusion at 10 mg/kg weekly (Cohort 1, 8 weeks) or 25 mg/kg bi-weekly (Cohort 2, 16 weeks).
  Other Names: dB4C7 mAb

SUMMARY:
The purpose of this phase II study is to evaluate the safety, tolerability and efficacy of two multi-dose regimens of UB-421 monotherapy in replacement of HAART in HIV-1 infected adults with virological suppression.

DETAILED DESCRIPTION:
This is an open-label, Phase II study to evaluate the safety, tolerability and efficacy of two multi-dose regimens of UB-421 monotherapy in replacement of HAART in HIV-1 infected adults with virological suppression. In this study, approximately 29 subjects will be enrolled to receive one of the two UB-421 regimens as the monotherapy in replacement of HARRT treatment. Subjects assigned to Cohort 1 will receive UB-421 infusion at 10 mg/kg weekly for 8 weeks; subjects assigned to Cohort 2 will receive UB-421 infusion at 25 mg/kg bi-weekly for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 sero-positive
* Aged 20 years or older
* Have received HAART treatment
* CD4+ T cell count ≧ 350 cells/mm3
* HIV-1 plasma RNA level remains below the limit of
* Were not breastfeeding for women
* Subjects with a negative serum pregnancy test result at screening visit for women of childbearing potential
* Subjects agree on using birth control barrier (female or male condom) during the entire study period
* Subjects sign the informed consent before undergoing any study procedures

Exclusion Criteria:

* Any active infection except for HIV, and required immediate therapy
* Any active AIDS-defining illness per Category B and Category C conditions according to the U.S. Centers for Disease Control and Prevention (CDC) Classification System for HIV Infection
* Any documented CD4+ T cell count < 200 cells/mm3 within the past 12 weeks before screening visit
* Any significant diseases (other than HIV-1 infection) or clinically significant findings, including psychiatric and behavioral problems, determined from screening, medical history, and/or physical examination that, in the investigator's opinion, would preclude the subject from participating in this study
* Any vaccination within 8 weeks prior to the first dose of study drug
* Any immunomodulating therapy (including interferon and steroid) or systemic chemotherapy within 12 weeks prior to the first dose of study drug
* Any illicit intravenous drugs within 12 weeks prior to the first dose of study drug
* Any current alcohol or illicit drug use that, in the investigator's opinion, will interfere with the subject's ability to comply with the dosing, visit schedules and protocol evaluations
* More than one change of HAART regimen because of virologic failure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 17 weeks for cohort 1, 25 weeks for cohort 2

SECONDARY OUTCOMES:
Peak concentration of UB-421 | 8 weeks for cohort 1, 15 weeks for cohort 2
Trough concentration of UB-421 | 8 weeks for cohort 1, 15 weeks for cohort 2

CONTACTS AND LOCATIONS:
Overall Officials: Wing Wai Wong, M.D., Principal Investigator — Taiwan, Taipei Veterans General Hospital; Yen Hsu Chen, M.D. PhD., Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital; Hung Chin Tsai, M.D. PhD., Principal Investigator — Taiwan, Kaohsiung Veterans General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Wang CY, Wong WW, Tsai HC, Chen YH, Kuo BS, Lynn S, Blazkova J, Clarridge KE, Su HW, Lin CY, Tseng FC, Lai A, Yang FH, Lin CH, Tseng W, Lin HY, Finstad CL, Wong-Staal F, Hanson CV, Chun TW, Liao MJ. Effect of Anti-CD4 Antibody UB-421 on HIV-1 Rebound after Treatment Interruption. N Engl J Med. 2019 Apr 18;380(16):1535-1545. doi: 10.1056/NEJMoa1802264. PMID 30995373